CLINICAL TRIAL: NCT04569604
Title: Impaired Quality of Life and Cognitive Function in Patients With Hypoparathyroidism Might be Explained by Disturbed Capillary Flow Patterns in the Brain
Brief Title: QoL and Cognitive Function in Patients With Hypoparathyroidism
Acronym: MR-hypoPT
Status: Completed | Type: Observational
Sponsor: University of Aarhus (Other)
Responsible Party: Principal Investigator, Tanja Sikjær, Principal Investigator, MD, PhD, University of Aarhus
Other Study IDs: #11102018; 1-10-72-304-18 (Other: Ethical Committee of The Central Denmark Region)
Record Dates: First submitted 2019-09-02; First posted 2020-09-30 (Actual); Last update posted 2021-12-23 (Actual); Status verified 2021-12

CONDITIONS: Hypoparathyroidism; Pseudo Hypoparathyroidism
Keywords: Quality of Life; MRI; Cognitive Impairment; Hypoparathyroidism; Pseudohypoparathyroidism
MeSH Terms: conditions — Hypoparathyroidism; Pseudohypoparathyroidism; Cognitive Dysfunction | interventions — Magnetic Resonance Imaging; Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Plasma, serum and 24hr urine samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Postsurgical hypoparathyroidism: Patients with hypoparathyroidism for 3 or more years after neck surgery
  Interventions: Diagnostic Test: MRI scans; Diagnostic Test: Neuro cognitive tests; Diagnostic Test: Questionnaires on Quality of Life; Diagnostic Test: Blood samples; Diagnostic Test: 24 hr urine samples
- Non-surgical hypoparathyroidism: Patients with hypoparathyroidism for 3 or more years without neck surgery
  Interventions: Diagnostic Test: MRI scans; Diagnostic Test: Neuro cognitive tests; Diagnostic Test: Questionnaires on Quality of Life; Diagnostic Test: Blood samples; Diagnostic Test: 24 hr urine samples
- Pseudohypoparathyroidism: Patients with the diagnosis of Pseudohypoparathyroidism
  Interventions: Diagnostic Test: MRI scans; Diagnostic Test: Neuro cognitive tests; Diagnostic Test: Questionnaires on Quality of Life; Diagnostic Test: Blood samples; Diagnostic Test: 24 hr urine samples
- Healthy controls: 25 controls from the background population matched on age (±3 years), gender and level of education with the 25 patients with postsurgical hypoparathyroidism
  Interventions: Diagnostic Test: MRI scans; Diagnostic Test: Neuro cognitive tests; Diagnostic Test: Questionnaires on Quality of Life; Diagnostic Test: Blood samples; Diagnostic Test: 24 hr urine samples

INTERVENTIONS:
Diagnostic Test: MRI scans — Contrast-enhanced, magnetic resonance imaging (MRI) based method to detect disturbances in microvascular flow patterns in the human brain
Diagnostic Test: Neuro cognitive tests — Standard neuropsychological test battery consists of validated tests to assess cognitive domains including verbal and visual memory, attention, language, visuospatial and executive functioning.
Diagnostic Test: Questionnaires on Quality of Life — SF36v2, WHO-5 well-being index, HPQ28, Symptom questionnaire, and a general questionnaire on background information, medication and diet.
Diagnostic Test: Blood samples — Markers of calcium homeostasis, inflammatory markers and hematology.
Diagnostic Test: 24 hr urine samples — 24 hr urine content of calcium, phosphate, magnesium, and creatinine.

SUMMARY:
Hypoparathyroidism (HypoPT) is a disease with inadequate production of parathyroid hormone (PTH) from the parathyroid glands leading to hypocalcemia. The most common form is postsurgical HypoPT due to neck surgery resulting in removed or damaged parathyroid glands.

HypoPT is a complex disease with a reduced Quality of life, mild cognitive impairment and in some patients have brain calcifications.

The aim of the present study is to investigate the cognitive function in patients with postsurgical and non-surgical (HypoPT) by neuropsychological assessments and magnetic resonance imaging (MRI).

The investigators will apply a contrast-enhanced MRI based method to HypoPT patients and age- and gender matched controls to examine whether capillary dysfunction can be detected, and whether symptom severity across patients correlates with the degree of capillary dysfunction in certain brain regions. To our knowledge there have been no previous studies on cognitive impairment and its origin in patients with HypoPT. The investigators hypothesize that the symptoms of HypoPT patients represent various degrees of capillary dysfunction, which interfere with their brain function.

DETAILED DESCRIPTION:
Hypoparathyroidism (HypoPT) is a disease with inadequate production of parathyroid hormone (PTH) from the parathyroid glands leading to hypocalcemia. The most common form is postsurgical HypoPT due to neck surgery resulting in removed or damaged parathyroid glands. Postsurgical HypoPT has a prevalence of 22/100,000 inhabitants in Denmark. Nonsurgical HypoPT is most often caused by mutations in different genes or on an autoimmune basis, the prevalence of nonsurgical HypoPT is 2.3/100,000 inhabitants in Denmark. If the gene mutation is within the GNAS gene or upstream of the GNAS complex locus it causes PseudoHypoPT (PHP), which is characterized by target organ resistance to PTH, also resulting in hypocalcaemia and hyperphosphatemia as in post- and nonsurgical HypoPT, but in this case with high or normal levels of plasma PTH. PHP is a very rare disease with a prevalence of 1/100,000 inhabitants in Denmark.

Others and the investigators have previously shown that HypoPT and/or hypocalcemia may affect quality of life (QoL). In most cases, severe symptoms and findings diminished or disappeared when plasma calcium levels are restored to normal, but as some of the above mentioned studies have shown, the reduced QoL is still present despite normal calcium levels. Symptoms are describes as minor cognitive impairment (MCI), with confusion, forgetfulness, and lack of focus and mental clarity. Another important finding in some of the patients with HypoPT is calcifications of the basal ganglia as described in several case reports, the knowledge of the origin and importance of these is so far limited. Patients with PHP have previously been described to have a higher risk of calcifications of the lens and subcutaneous calcifications, and therefore might also be at higher risk of calcifications in the brain.

The oxygen availability in brain tissue is traditionally thought to depend on regional cerebral blood flow (CBF). Accordingly, brain oxygenation is only expected to impair brain function in cases where CBF is critically reduced, cerebral ischemia. This paradigm was recently shown to be in error: While CBF determines the oxygen supply, the microscopic distribution of blood flows across the capillary bed determines the extent to which this oxygen can be extracted by the tissue. In fact, capillary flow patterns can become so disturbed that the metabolic needs of brain function and survival can no longer be met - although CBF remains inconspicuous. Capillary dysfunction denotes this overlooked source of hypoxia: A state in which capillary flow patterns cannot homogenize, giving rise to tissue hypoxia, oxidative stress, local inflammation, and - if severe - long-term neurodegeneration. The investigators hypothesize that the symptoms of HypoPT patients represent various degrees of capillary dysfunction, which interfere with their brain function.

The purpose of the study is to investigate whether HypoPT patients are affected by capillary dysfunction, a condition in which capillary flow disturbances interfere with brain oxygenation.

The hypothesis derives from findings that cerebral calcifications similar to those found in HypoPT are observed in familial idiopathic basal ganglia calcification (IBGC), which is a disease of cerebral pericytes. Pericytes are localized in the basement membrane of capillaries, where they maintain blood brain barrier (BBB) function and - in close interaction with endothelial cells - basement membrane and capillary wall integrity. They are contractile and take part in blood flow regulation. They control the trafficking of immune cells across the vessel wall and possess stem/progenitor cell functions. As such, they play a key role in tissue repair, scarring, and fibrosis, and along with endothelial cells, they seemingly have the potential to become bone-forming cells.

Pericytes (now referred to as 'mural cells') are characterized by several membrane proteins, one of which (SLC9A3R1 - solute carrier family 9, isoform A3, regulatory factor 1, also known as EBP50, NHERF) binds to parathyroid hormone 1 receptor (PTH1R) on one hand, and to plasma derived growth factor (PDGF) receptor β (PDGFβ) on the other, potentiating its activity. The physiological role of these receptors is poorly understood. Receptors for PTH and Parathyroid hormone-related protein (PTH-rP) have been observed in both pericytes and smooth muscle cells of various tissue types, while PTH-rP is expressed in the endothelium, acting as a vasodilator. There is hence reason to believe that the function of capillary pericytes - and hence capillary flow patterns - could be altered in HypoPT.

The investigators have developed a contrast-enhanced, magnetic resonance imaging (MRI) based method to detect disturbances in microvascular flow patterns in the human brain and demonstrated that knowledge of these flow patterns - as indexed by the capillary transit-time heterogeneity (CTH) - allow us to better predict oxygen extraction efficacy as determined by a gold-standard positron emission tomography (PET). The investigators have now found abnormal microvascular flow patterns in patients with Alzheimer's disease (AD) or mild cognitive impairment (MCI) compared to healthy, age-matched controls without cardiovascular risk factors, and demonstrated that the degree of capillary dysfunction correlated with their cognitive impairment. The investigators found a similar correlation in another AD patient cohort, and most recently detected capillary dysfunction in patients with late-onset depression compared to controls. In view of these findings, and the similarity between the symptomatology of HypoPT and depression, the investigators now propose to apply our MRI method to HypoPT patients and age- and gender matched controls to examine whether capillary dysfunction can be detected, and whether symptom severity across patients correlates with the degree of capillary dysfunction in certain brain regions.

The aim is to investigate the cognitive function in patients with postsurgical, non-surgical and pseudoHypoPT by neuropsychological assessments and MRI. The contrast-enhanced MRI based method will be applied to HypoPT patients and age- and gender matched controls to examine whether capillary dysfunction can be detected, and whether symptom severity across patients correlates with the degree of capillary dysfunction in certain brain regions.

The investigators hypothesize that the symptoms of HypoPT patients represent various degrees of capillary dysfunction, which interfere with their brain function.

Methods:

MRI scans: The investigators plan to acquire the following MRI sequences:

1. Dynamic susceptibility contrast perfusion MRI will be applied for measurement of capillary function and regional blood flow and volume as estimated by our by parametric approach.
2. For further characterization of the microcirculation, resting state functional MRI will be acquired. This sequence can be acquired in combination with the perfusion scan and thus requires very little extra scanning time.
3. Fluid attenuated inversion recovery (FLAIR) images will be acquired for estimation of white matter hyperintensities (WMH) and possible subcortical infarcts or lacunas.
4. A fast diffusion kurtosis imaging (DKI) sequence will be applied for estimation of microstructural integrity of gray and white matter (e.g. dendrite density and white matter tract integrity).
5. T1-weighted MRI will be utilized for accurate morphological characterization of cerebral structures, such as hippocampus, basal ganglia, cortex and major tracts. In addition, the high-resolution images enable accurate mapping of the functional data (perfusion, fMRI, DKI).

Neuropsychological testing (NPT): The standard neuropsychological test battery consists of validated tests to assess cognitive domains including verbal and visual memory, attention, language, visuospatial and executive functioning.

Cognitive batteries: Cogstate battery for assessing cognitive function in adults with mild cognitive impairment (MCI). The tests used are D-KEFS: TrailMaking A and B, Verbal Fluency Test, and Color-Word Interference Test. The WAIS-IV: Coding, Symbol search, Digit span, and Arithmetic. The BVMT-R: delayed recall and total learning. Lastly the RAVLT: delayed recall and total learning.

Questionnaires: SF36v2, WHO-5 well-being index, Symptom questionnaire, and a general questionnaire on background information, medication and diet, and HPQ28.

Biochemistry: Ionized calcium, PTH, phosphate, magnesium, eGFR, creatinine, High sensitive CRP, 25-hydroxyvitamin D, calcitriol, and white blood cell count. Neuroinflammation and systemic inflammatory markers (pro-inflammatory cytokines), and 24-hr urine.

Statistical Analysis Plan: Group difference will be examined using student T test for continuous variables and Pearsons X^2 test for categorical variables. Statistical maps of differences in perfusion parameters between patients and controls will be calculated at each surface vertex using a vertex specific general linear model with cortical thickness, white matter hyperintensity load ((WMHL) given as percentage white matter hyperintensities volume of whole brain volume)), age, and gender as covariates. The investigators will add cortical thickness as covariate to account for any systematic effects of cortical thickness on the perfusion measurements, such as partial volume effects. All statistical maps will be thresholded at p=0.05 (uncorrected and corrected). All statistical tests for the MRI scans are carried out using R version 3.2.2 (The R Foundation for Statistical Computing) and SPM12 (Wellcome Trust Centre for Neuroimaging) running on Matlab R2016a (MathWorks Inc). Other statistical test will be carried out by SPSS 24 (IBM, USA) Justification for sample size: In a previous study by Eskildsen et al. the contrast-enhanced MRI based method has been applied to 18 patients with Alzheimer's disease or MCI compared to 19 healthy, age-matched controls without cardiovascular risk factors and it demonstrated that the degree of capillary dysfunction correlated with their cognitive impairment. The investigators found a similar correlation in another patient cohort with Alzheimer's disease, and most recently detected capillary dysfunction in patients with late-onset depression compared to controls. Taking the above mentioned results and the sizes of the cohorts in consideration, the investigators have estimated that our sample size is enough to show if there is a correlation between cognitive impairment measured by neuropsychological assessment and capillary transit time heterogeneity.

Safety and ethnical evaluations: The investigators will follow the standard operating procedures regarding contrast enhanced MRI scans. Peripheral venous catheter will be used for administration of PET tracers and MRI contrast. It can result in mild local pain and a hematoma. The risk of infection is negligible. There are no known risks (neither short- nor long-term) related to MRI. Gadolinium-chelate (Gd) contrast is used. The standard dose of gadolinium (Gd)-containing MRI-contrast is 0.1 mmol/kg, but in this study there will be used up to 0.3 mmol/kg.

Perspectives: If successful and study findings provides a basis for improved understanding of cognitive symptoms in HypoPT, further investigations on effects of PTH replacement therapy on investigated indices should be considered. A future project could be performing the MRI scan before and after injection of PTH to determine whether a change in capillary transit time heterogeneity could be detected.

ELIGIBILITY:
Inclusion Criteria:

* Patients:
* Male or female with age between 18 and 70 years.
* A low endogenous PTH production as verified by low plasma levels of intact PTH, necessitating treatment with 1-αhydroxylated vitamin D analogs.
* HypoPT for 3 years with continuous alphacalcidol or calcitriol treatment prior to study entry (except for the patients with PHP).
* Stable P-calcium levels 1 month prior to inclusion.
* In case of thyroid disease, TSH within reference range within the last year
* Speaks and reads Danish

Controls:

* Male or female with age between 18 and 80 years.
* No known diseases in the calcium homeostasis
* Speaks and reads Danish

Exclusion Criteria:

* Reduced kidney function (eGFR < 30 mL/min/1.73m2).
* Diabetes type 1 or 2
* History of hypertension for more than two years (treated or untreated)
* Clinical suspicion of major depression (also if treated)
* Clinical suspicion of alcohol-related dementia
* Other organic or psychiatric cause the patients symptoms
* Contraindications to contrast-enhanced MRI.
* Metal implants close to the head, which will interfere with the MRI or pacemaker. The patients will complete a metal scheme.
* Claustrophobia
* Unwillingness to participate

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The patients with postsurgical, non-surgical and pseudo hypoparathyroidism will be invited from our outpatient clinic to participate in the study.
  The healthy controls will be randomly recruited from the background population by an extract from the CPR register and an invitation to participate in the study will be send by electronic letter.
Sampling Method: Non-Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Capillary transit time heterogeneity | MRI scan performed at baseline, no follow-up up. It takes 1 hour to perform
  Capillary transit time heterogeneity is measured by MRI scans

SECONDARY OUTCOMES:
Index 1: Processing speed | Neuropsychological tests are performed immediately before or immediately after the MRI scan and scheduled to take 1½ hours.
  Index 1 consist of the following tests
  1. Coding (WAIS-IV) scaled score
  2. Symbol search (WIAS-IV) scaled score
  A composit score from the above tests will be calculated and compared to the control group and normative data.
Index 2: Working memory | Neuropsychological tests are performed immediately before or immediately after the MRI scan and scheduled to take 1½ hours.
  Index 2 consist of the following tests
  1. Digit span (WAIS-IV) scaled score
  2. Arithmetic (WAIS-IV) scaled score
  A composit score will be calculated from the above tests and compared to the control group and normative data.
Index 3: Executive function | Neuropsychological tests are performed immediately before or immediately after the MRI scan and scheduled to take 1½ hours.
  Index 3 consist of the following tests
  1. Trail Making Test (D-KEFS) scaled score
  2. Verbal Fluency Test (D-KEFS) scaled score
  3. Color-Word Interference Test (D-KEFS) scaled score
  A composit score will be calculated from the above tests and compared to the control group and normative data.
Index 4: Verbal learning and memory | Neuropsychological tests are performed immediately before or immediately after the MRI scan and scheduled to take 1½ hours.
  Index 4 consist of the following tests
  1. Rey Auditory Verbal Learning Test (RAVLT) total learning scaled score
  2. Rey Auditory Verbal Learning Test (RAVLT) delayed recall scaled score
  A composit score will be calculated from the above tests and compared to the control group and normative data.
Index 5: Visual learning and memory | Neuropsychological tests are performed immediately before or immediately after the MRI scan and scheduled to take 1½ hours.
  Index 4 consist of the following tests
  1. Brief Visuospatial Memory Test-Revised (BVMT-R) total learning scaled score
  2. Brief Visuospatial Memory Test-Revised (BVMT-R) delayed recall scaled score
  A composit score will be calculated from the above tests and compared to the control group and normative data.
Correlation of calcifications in the brain and cognitive function. | The MRI scan: Baseline visit (duration 1 hr.). Neuropsychological tests are performed immediately before or immidiatly after the MRI.The analyses of the calcifications: Three months after the last subject has finished the study ( duration 1-2 mo)
  Calcifications:
  The calcifications will be visually inspected on the PETRA sequense of the MRI scans.
  It will defined by its location (Globus pallidus, Thalamus, caudate nucleus, cortex, putamen, or cerebellum) and then defined in accordance with its size as listed below:
  The calcifications are going to be divided into 4 categories according to size:
  1. "barely recognizable" / up to approx. 1 mm,
  2. "small" / up to approx. 3 mm,
  3. "medium" / up to approx. 8 mm,
  4. "large" / approx. > 8 mm. The size classification will be based on segmentation of the calcification finding the maximum cross section measured.
  The most severe score will be attributed if more than one calcification is present in one location.
  The calcifikation load of the patient will be an addition of scores from the different locations.
  There will be tested for a correlation of the calcification load and the scores from the Index 1, 2, 3, 4, and 5 of the neuropsychological tests.
Difference in capillary transit time heterogeneity between patients and healthy controls | MRI scan performed at baseline, no follow-up up. It takes 1 hour to perform
  Capillary transit time heterogeneity is measured by MRI scans and compared between groups
Difference in Quality of Life between patients and healthy controls. | The questionnaires were completed online within 3 weeks after the day with the MRI scand and the neurocognitive testing.
  Quality of life is measured by three different questionnaires.
  1. 36-Item Short Form Survey version 2 (SF36v2): A questionnaire with 36 questions on mental and physical complaints. The higher score, the better.
  2. : The WHO-5 wellbeing index: 5 questions on well being. The higher score the better.
  3. HPQ-28: A disease specific questionnaire designed for patients with Hypoparathyriodsm. The lower the score the better.

CONTACTS AND LOCATIONS:
Overall Officials: Tanja T Sikjær, MD, PhD, Principal Investigator — Department of Endocrinology and Internal Medicine, Aarhus University Hospital
Locations (1):
- Clinic for Osteoporosis, Aarhus University Hospital, Aarhus N, Jutland, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Underbjerg L, Sikjaer T, Mosekilde L, Rejnmark L. Cardiovascular and renal complications to postsurgical hypoparathyroidism: a Danish nationwide controlled historic follow-up study. J Bone Miner Res. 2013 Nov;28(11):2277-85. doi: 10.1002/jbmr.1979. PMID 23661265
- [Background] Underbjerg L, Sikjaer T, Mosekilde L, Rejnmark L. The Epidemiology of Nonsurgical Hypoparathyroidism in Denmark: A Nationwide Case Finding Study. J Bone Miner Res. 2015 Sep;30(9):1738-44. doi: 10.1002/jbmr.2501. Epub 2015 May 31. PMID 25753591
- [Background] Underbjerg L, Sikjaer T, Mosekilde L, Rejnmark L. Pseudohypoparathyroidism - epidemiology, mortality and risk of complications. Clin Endocrinol (Oxf). 2016 Jun;84(6):904-11. doi: 10.1111/cen.12948. Epub 2015 Oct 19. PMID 26387561
- [Background] Bohrer T, Krannich JH. Depression as a manifestation of latent chronic hypoparathyroidism. World J Biol Psychiatry. 2007;8(1):56-9. doi: 10.1080/15622970600995146. PMID 17366354
- [Background] Lawlor BA. Hypocalcemia, hypoparathyroidism, and organic anxiety syndrome. J Clin Psychiatry. 1988 Aug;49(8):317-8. PMID 3045102
- [Background] Snowdon JA, Macfie AC, Pearce JB. Hypocalcaemic myopathy with paranoid psychosis. J Neurol Neurosurg Psychiatry. 1976 Jan;39(1):48-52. doi: 10.1136/jnnp.39.1.48. PMID 1255212
- [Background] Arlt W, Fremerey C, Callies F, Reincke M, Schneider P, Timmermann W, Allolio B. Well-being, mood and calcium homeostasis in patients with hypoparathyroidism receiving standard treatment with calcium and vitamin D. Eur J Endocrinol. 2002 Feb;146(2):215-22. doi: 10.1530/eje.0.1460215. PMID 11834431
- [Background] Astor MC, Lovas K, Debowska A, Eriksen EF, Evang JA, Fossum C, Fougner KJ, Holte SE, Lima K, Moe RB, Myhre AG, Kemp EH, Nedrebo BG, Svartberg J, Husebye ES. Epidemiology and Health-Related Quality of Life in Hypoparathyroidism in Norway. J Clin Endocrinol Metab. 2016 Aug;101(8):3045-53. doi: 10.1210/jc.2016-1477. Epub 2016 May 17. PMID 27186861
- [Background] Sikjaer T, Moser E, Rolighed L, Underbjerg L, Bislev LS, Mosekilde L, Rejnmark L. Concurrent Hypoparathyroidism Is Associated With Impaired Physical Function and Quality of Life in Hypothyroidism. J Bone Miner Res. 2016 Jul;31(7):1440-8. doi: 10.1002/jbmr.2812. Epub 2016 Mar 31. PMID 26865527
- [Background] Sikjaer T, Rolighed L, Hess A, Fuglsang-Frederiksen A, Mosekilde L, Rejnmark L. Effects of PTH(1-84) therapy on muscle function and quality of life in hypoparathyroidism: results from a randomized controlled trial. Osteoporos Int. 2014 Jun;25(6):1717-26. doi: 10.1007/s00198-014-2677-6. Epub 2014 Apr 1. PMID 24687385
- [Background] Velasco PJ, Manshadi M, Breen K, Lippmann S. Psychiatric aspects of parathyroid disease. Psychosomatics. 1999 Nov-Dec;40(6):486-90. doi: 10.1016/s0033-3182(99)71186-2. PMID 10581976
- [Background] Underbjerg L, Sikjaer T, Rejnmark L. Health-related quality of life in patients with nonsurgical hypoparathyroidism and pseudohypoparathyroidism. Clin Endocrinol (Oxf). 2018 Jun;88(6):838-847. doi: 10.1111/cen.13593. Epub 2018 Apr 3. PMID 29520810
- [Background] Abiusi G, Dominguez RO, Parada Marcilla M, Lesyk S, Laguarde N, Yobstraibizer F. [Asymptomatic encephalic calcifications in postsurgical hypoparathyroidism]. Neurologia. 2009 Sep;24(7):454-6. Spanish. PMID 19921554
- [Background] Basak RC. A case report of Basal Ganglia calcification - a rare finding of hypoparathyroidism. Oman Med J. 2009 Jul;24(3):220-2. doi: 10.5001/omj.2009.44. PMID 22224190
- [Background] Bhimani S, Sarwar M, Virapongse C, Rojas R, Freilich M. Computed tomography of cerebrovascular calcifications in postsurgical hypoparathyroidism. J Comput Assist Tomogr. 1985 Jan-Feb;9(1):121-4. doi: 10.1097/00004728-198501000-00022. PMID 3968258
- [Background] Chow KS, Lu DN. [Primary hypoparathyroidism with basal ganglia calcification: report of a case]. Zhonghua Min Guo Xiao Er Ke Yi Xue Hui Za Zhi. 1989 Mar-Apr;30(2):129-33. Chinese. PMID 2637591
- [Background] DANOWSKI TS, LASSER EC, WECHSLER RL. Calcification of basal ganglia in post-thyroidectomy hypoparathyroidism. Metabolism. 1960 Nov;9:1064-5. No abstract available. PMID 13719679
- [Background] EATON, L. M. & HAINES, S. F. Parathyroid insuffiency with symmetrical cerebral calcification. Journal of the American Medical Association 113, 749-753 (1939).
- [Background] Forman MB, Sandler MP, Danziger A, Kalk WJ. Basal ganglia calcification in postoperative hypoparathyroidism. Clin Endocrinol (Oxf). 1980 Apr;12(4):385-90. doi: 10.1111/j.1365-2265.1980.tb02725.x. PMID 7379319
- [Background] Fukunaga M, Otsuka N, Ono S, Kajihara Y, Nishishita S, Nakano Y, Yamamoto I, Torizuka K, Morita R. Computed tomography of basal ganglia calcifications in pseudo- and idiopathic hypoparathyroidism. Radiat Med. 1987 Nov-Dec;5(6):187-90. PMID 3452848
- [Background] Garcia Urra D, Barquero Jimenez MS, Varela de Seijas E, Rico Lenza H. [Calcification of the basal ganglia and hypoparathyroidism: Fahr disease. Study of a family]. Arch Neurobiol (Madr). 1990 Jan-Feb;53(1):18-22. Spanish. PMID 2393337
- [Background] Goncalves Junior JC, Oliveira TS, Arantes HP, Goncalves FT, Fonseca AR, Jorge PT. [Cerebral calcifications due to hypoparathyroidism: considerations about cases diagnosed many years after partial thyroidectomy]. Arq Bras Endocrinol Metabol. 2006 Dec;50(6):1133-7. doi: 10.1590/s0004-27302006000600023. Portuguese. PMID 17221123
- [Background] Jorens PG, Appel BJ, Hilte FA, Mahler C, De Deyn PP. Basal ganglia calcifications in postoperative hypoparathyroidism: a case with unusual characteristics. Acta Neurol Scand. 1991 Feb;83(2):137-40. doi: 10.1111/j.1600-0404.1991.tb04663.x. PMID 1902012
- [Background] Jorgensen H, Vogt H. [Familial, idiopathic hypoparathyroidism with intracerebral calcifications and extrapyramidal symptoms]. Tidsskr Nor Laegeforen. 1977 May 30;97(15):771-4. No abstract available. Norwegian. PMID 194354
- [Background] Karimi M, Rasekhi AR, Rasekh M, Nabavizadeh SA, Assadsangabi R, Amirhakimi GH. Hypoparathyroidism and intracerebral calcification in patients with beta-thalassemia major. Eur J Radiol. 2009 Jun;70(3):481-4. doi: 10.1016/j.ejrad.2008.02.003. Epub 2008 Mar 25. PMID 18367361
- [Background] Mahmoodi M, De Sanctis V, Karimi M. Diffuse intracerebral calcification in a beta-thalassaemia major patient with hypoparathyroidism: a case report. Pediatr Endocrinol Rev. 2011 Mar;8 Suppl 2:331-3. PMID 21705988
- [Background] Kartin P, Zupevc M, Pogacnik T, Cerk M. Calcification of basal ganglia, postoperative hypoparathyroidism and extrapyramidal, cerebellar, pyramidal motor manifestations. J Neurol. 1982;227(3):171-6. doi: 10.1007/BF00313572. PMID 6181225
- [Background] LEVIN P. Intracranial calcification associated with hypoparathyroidism. Bull N Y Acad Med. 1962 Sep;38(9):632-7. No abstract available. PMID 14464573
- [Background] Polverosi R, Zambelli C, Sbeghen R. [Calcification of the basal nuclei in hypoparathyroidism. The computed and magnetic resonance tomographic aspects]. Radiol Med. 1994 Jan-Feb;87(1-2):12-5. Italian. PMID 8128014
- [Background] Preusser M, Kitzwoegerer M, Budka H, Brugger S. Bilateral striopallidodentate calcification (Fahr's syndrome) and multiple system atrophy in a patient with longstanding hypoparathyroidism. Neuropathology. 2007 Oct;27(5):453-6. doi: 10.1111/j.1440-1789.2007.00790.x. PMID 18018479
- [Background] Rastogi R, Beauchamp NJ, Ladenson PW. Calcification of the basal ganglia in chronic hypoparathyroidism. J Clin Endocrinol Metab. 2003 Apr;88(4):1476-7. doi: 10.1210/jc.2002-021804. No abstract available. PMID 12679425
- [Background] Stelmasiak Z, Tarach JS, Nowicka-Tarach BM, Mitosek-Szewczyk K, Drop A. Idiopathic hypoparathyroidism with intracranial calcifications and dominant skin manifestations. Med Sci Monit. 2000 Jan-Feb;6(1):145-50. PMID 11208303
- [Background] Levine MA. Pseudohypoparathyroidism: from bedside to bench and back. J Bone Miner Res. 1999 Aug;14(8):1255-60. doi: 10.1359/jbmr.1999.14.8.1255. No abstract available. PMID 10457257
- [Background] Mantovani G, Bastepe M, Monk D, de Sanctis L, Thiele S, Usardi A, Ahmed SF, Bufo R, Choplin T, De Filippo G, Devernois G, Eggermann T, Elli FM, Freson K, Garcia Ramirez A, Germain-Lee EL, Groussin L, Hamdy N, Hanna P, Hiort O, Juppner H, Kamenicky P, Knight N, Kottler ML, Le Norcy E, Lecumberri B, Levine MA, Makitie O, Martin R, Martos-Moreno GA, Minagawa M, Murray P, Pereda A, Pignolo R, Rejnmark L, Rodado R, Rothenbuhler A, Saraff V, Shoemaker AH, Shore EM, Silve C, Turan S, Woods P, Zillikens MC, Perez de Nanclares G, Linglart A. Diagnosis and management of pseudohypoparathyroidism and related disorders: first international Consensus Statement. Nat Rev Endocrinol. 2018 Aug;14(8):476-500. doi: 10.1038/s41574-018-0042-0. PMID 29959430
- [Background] Jespersen SN, Ostergaard L. The roles of cerebral blood flow, capillary transit time heterogeneity, and oxygen tension in brain oxygenation and metabolism. J Cereb Blood Flow Metab. 2012 Feb;32(2):264-77. doi: 10.1038/jcbfm.2011.153. Epub 2011 Nov 2. PMID 22044867
- [Background] Ostergaard L, Jespersen SN, Mouridsen K, Mikkelsen IK, Jonsdottir KY, Tietze A, Blicher JU, Aamand R, Hjort N, Iversen NK, Cai C, Hougaard KD, Simonsen CZ, Von Weitzel-Mudersbach P, Modrau B, Nagenthiraja K, Riisgaard Ribe L, Hansen MB, Bekke SL, Dahlman MG, Puig J, Pedraza S, Serena J, Cho TH, Siemonsen S, Thomalla G, Fiehler J, Nighoghossian N, Andersen G. The role of the cerebral capillaries in acute ischemic stroke: the extended penumbra model. J Cereb Blood Flow Metab. 2013 May;33(5):635-48. doi: 10.1038/jcbfm.2013.18. Epub 2013 Feb 27. PMID 23443173
- [Background] Betsholtz C, Keller A. PDGF, pericytes and the pathogenesis of idiopathic basal ganglia calcification (IBGC). Brain Pathol. 2014 Jul;24(4):387-95. doi: 10.1111/bpa.12158. PMID 24946076
- [Background] Armulik A, Genove G, Mae M, Nisancioglu MH, Wallgard E, Niaudet C, He L, Norlin J, Lindblom P, Strittmatter K, Johansson BR, Betsholtz C. Pericytes regulate the blood-brain barrier. Nature. 2010 Nov 25;468(7323):557-61. doi: 10.1038/nature09522. Epub 2010 Oct 13. PMID 20944627
- [Background] Armulik A, Abramsson A, Betsholtz C. Endothelial/pericyte interactions. Circ Res. 2005 Sep 16;97(6):512-23. doi: 10.1161/01.RES.0000182903.16652.d7. PMID 16166562
- [Background] Hall CN, Reynell C, Gesslein B, Hamilton NB, Mishra A, Sutherland BA, O'Farrell FM, Buchan AM, Lauritzen M, Attwell D. Capillary pericytes regulate cerebral blood flow in health and disease. Nature. 2014 Apr 3;508(7494):55-60. doi: 10.1038/nature13165. Epub 2014 Mar 26. PMID 24670647
- [Background] Funk JL, Wei H, Downey KJ, Yocum D, Benjamin JB, Carley W. Expression of PTHrP and its cognate receptor in the rheumatoid synovial microcirculation. Biochem Biophys Res Commun. 2002 Oct 4;297(4):890-7. doi: 10.1016/s0006-291x(02)02263-5. PMID 12359237
- [Background] Mouridsen K, Hansen MB, Ostergaard L, Jespersen SN. Reliable estimation of capillary transit time distributions using DSC-MRI. J Cereb Blood Flow Metab. 2014 Sep;34(9):1511-21. doi: 10.1038/jcbfm.2014.111. Epub 2014 Jun 18. PMID 24938401
- [Background] Mouridsen K, Friston K, Hjort N, Gyldensted L, Ostergaard L, Kiebel S. Bayesian estimation of cerebral perfusion using a physiological model of microvasculature. Neuroimage. 2006 Nov 1;33(2):570-9. doi: 10.1016/j.neuroimage.2006.06.015. Epub 2006 Sep 12. PMID 16971140
- [Background] Ostergaard L, Jespersen SN, Engedahl T, Gutierrez Jimenez E, Ashkanian M, Hansen MB, Eskildsen S, Mouridsen K. Capillary dysfunction: its detection and causative role in dementias and stroke. Curr Neurol Neurosci Rep. 2015 Jun;15(6):37. doi: 10.1007/s11910-015-0557-x. PMID 25956993
- [Background] Eskildsen SF, Gyldensted L, Nagenthiraja K, Nielsen RB, Hansen MB, Dalby RB, Frandsen J, Rodell A, Gyldensted C, Jespersen SN, Lund TE, Mouridsen K, Braendgaard H, Ostergaard L. Increased cortical capillary transit time heterogeneity in Alzheimer's disease: a DSC-MRI perfusion study. Neurobiol Aging. 2017 Feb;50:107-118. doi: 10.1016/j.neurobiolaging.2016.11.004. Epub 2016 Nov 19. PMID 27951412
- [Background] Nielsen RB, Egefjord L, Angleys H, Mouridsen K, Gejl M, Moller A, Brock B, Braendgaard H, Gottrup H, Rungby J, Eskildsen SF, Ostergaard L. Capillary dysfunction is associated with symptom severity and neurodegeneration in Alzheimer's disease. Alzheimers Dement. 2017 Oct;13(10):1143-1153. doi: 10.1016/j.jalz.2017.02.007. Epub 2017 Mar 23. PMID 28343848
- [Background] Mouridsen K, Christensen S, Gyldensted L, Ostergaard L. Automatic selection of arterial input function using cluster analysis. Magn Reson Med. 2006 Mar;55(3):524-31. doi: 10.1002/mrm.20759. PMID 16453314
- [Background] Hansen B, Khan AR, Shemesh N, Lund TE, Sangill R, Eskildsen SF, Ostergaard L, Jespersen SN. White matter biomarkers from fast protocols using axially symmetric diffusion kurtosis imaging. NMR Biomed. 2017 Sep;30(9):10.1002/nbm.3741. doi: 10.1002/nbm.3741. Epub 2017 May 22. PMID 28543843
- [Background] Hansen B, Lund TE, Sangill R, Jespersen SN. Experimentally and computationally fast method for estimation of a mean kurtosis. Magn Reson Med. 2013 Jun;69(6):1754-60. doi: 10.1002/mrm.24743. Epub 2013 Apr 15. PMID 23589312
- [Background] Hansen B, Shemesh N, Jespersen SN. Fast imaging of mean, axial and radial diffusion kurtosis. Neuroimage. 2016 Nov 15;142:381-393. doi: 10.1016/j.neuroimage.2016.08.022. Epub 2016 Aug 15. PMID 27539807
- [Background] Lewis, M. et al. Assessment of cognition in an adolescent Indigenous population. Australian Psychologist 45, 123-131, doi:10.1080/00050060903352998 (2010).
- [Background] Reitan, R. M. Validity of the Trail Making Test as an indicator of organic brain damage. Perceptual and Motor Skills 8 (1958).
- [Background] Wechsler, D. Wechsler Adult Intelligence Scale. Third edn, (The Psychological Corporation, 1997).
- [Background] Meyers, J. E. & Meyers, K. R. Rey Complex Figure Test and Recognition Trail. (Psychological Assessment Resources, 1995).
- [Background] Nielsen H, Knudsen L, Daugbjerg O. Normative data for eight neuropsychological tests based on a Danish sample. Scand J Psychol. 1989;30(1):37-45. doi: 10.1111/j.1467-9450.1989.tb01066.x. PMID 2740854
- [Background] Wilde D, Wilken L, Stamm B, Blaschke M, Heppner C, Chavanon ML, Leha A, Herrmann-Lingen C, Siggelkow H. The HPQ-Development and First Administration of a Questionnaire for Hypoparathyroid Patients. JBMR Plus. 2019 Nov 7;4(1):e10245. doi: 10.1002/jbm4.10245. eCollection 2020 Jan. PMID 31956849